CLINICAL TRIAL: NCT05002894
Title: Effect of Pilates Exercises On Fatigue In Post Menopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mohamed Nabil Hussein, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pilates Effect On Fatigue
Record Dates: First submitted 2021-07-01; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Fatigue
Keywords: fatigue; sleep disturbance
MeSH Terms: conditions — Fatigue; Parasomnias | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise group (Experimental): This group included twenty six post-menopausal women. They will participate in Pilates exercise, medical standard care for fatigue and advices to deal with fatigue. The Pilates exercises consisted of a set of 10 movements: bridging; hundred; roll up; one leg circle (both ways); single straight leg stretch; single leg kick; side kick up and down; side kick circles; rest position (stretch and relaxation); and curling ,women were instructed to perform 30 min per session, 3 sessions per week, for 8 weeks.
  Interventions: Other: Pilates exercises; Dietary Supplement: medical standard care for fatigue
- standard care group (Experimental): Each post-menopausal woman in both groups will receive a medical standard care for post-menopausal fatigue.
  Interventions: Dietary Supplement: medical standard care for fatigue

INTERVENTIONS:
Other: Pilates exercises — Pilates exercises for flexibility and stability
  Arms: exercise group
Dietary Supplement: medical standard care for fatigue — supplements and medical care

SUMMARY:
Pilates is a system of exercises using special apparatus, designed to improve physical strength, flexibility, and enhance mental awareness. Regular exercise of post-menopausal women has benefits of increased cardio-respiratory fitness, increased muscle strength and endurance, reduced body fatigue, improved morale, and increased ability to perform daily tasks with greater force.Thus the main objective of regular exercise is prevention of physical deterioration and optimizing functional capacity to improve overall postmenopausal women's quality of life.

DETAILED DESCRIPTION:
Fatigue has a negative impact on quality of life of postmenopausal women. Fatigue can be an overwhelming experience impacting the physical, emotional and social aspects of them. Fatigue can prevent them from carrying out their usual activities of daily living ,Menopause-related fatigue can be caused by changing estrogen levels, but it is often compounded by common symptoms, chief symptoms among these are vasomotor symptoms, which are experienced by up to 80% of women and include hot flashes and night sweats that can disrupt sleep , Pilates exercise considered a complementary therapy to treat fatigue in postmenopausal women. Pilates exercises are a healthy and effective method for improving the functional capacity, flexibility, fatigue, depression and quality of life of post menopause women ,They include stretching and strengthening exercises with controlled and precise movements that have indicated both mental and physical effects on post-menopausal women healthThe purpose of physical training using Pilates is to improve body functioning based on core strengthening that include rectus abdomens, transverse abdomen, erector spine, diaphragm and pelvic floor muscles. The six basic principles of Pilates exercise are centralization, concentration, control, precision, respiration and flow .

ELIGIBILITY:
Inclusion Criteria:

. All participants will be sedentary.

* All participants' ages will be ranged from 50-55 years.
* All participants body mass index will not exceed 30 kg/m2.
* All participants will be medically stable.
* All participants will be able to ambulate independently.
* All participants suffering from fatigue, when assessed with fatigue assessment scale (FAS) their scores should be >22.

Exclusion Criteria:

* • Post-menopausal women who have Uncontrolled hypertension.

  * Post-menopausal women who have Thyroid gland disorders.
  * Post-menopausal women who have History of syncope or arrhythmia induced by physical exercise.
  * Postmenopausal women who have any mental, neurological, vestibular, cardiovascular disorders or metabolic disease.
  * Postmenopausal women whose visual or hearing impairment did not allow possibility of intervention.
  * Postmenopausal women who have been received hormonal replacement therapy or any drug known to affect their physical activity.
  * Post-menopausal women who have any other problems that make it impossible to perform physical exercises.

Ages: 50 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 52 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
change in Fatigue Assessment Scale | immediately before the intervention (baseline value) and after 8 weeks of intervention
  Assess fatigue for postmenopausal women The total score ranges from 10 to 50.
  * A total FAS score < 22 indicates no fatigue.
  * A score ≥ 22 indicates fatigue

SECONDARY OUTCOMES:
change in Intreluken-6 test | immediately before the intervention (baseline value) and after 8 weeks of intervention
  Evaluate fatigue in post menopausal women it is a blood analysis It's normal range is 0-16.4 pg/mL
  Values higher than 16.4 indicate fatigue

OTHER OUTCOMES:
change in Pittsburgh Sleep Quality Index | immediately before the intervention (base line value) and after 8 weeks of intervention
  Self-report questionnaire that assesses sleep quality The scores range from 0 to 21, a score >5 be considered as a significant sleep disturbance.